CLINICAL TRIAL: NCT00440310
Title: A Multicenter Multinational Phase 3 Randomized Study to Evaluate the Safety and Efficacy of Treating Colorectal Cancer Patients With Recurrent Liver Metastases Using the Litx™ System Plus Chemotherapy as Compared to Chemotherapy Only
Brief Title: Phase 3 Trial of Litx™ Plus Chemotherapy vs. Chemotherapy Only Treating Colorectal Cancer Patients With Recurrent Liver Metastases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Light Sciences Oncology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LSO-OL006
Record Dates: First submitted 2007-02-23; First posted 2007-02-27 (Estimated); Results first posted 2015-08-25 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-07

CONDITIONS: Liver Metastases; Colorectal Neoplasms; Neoplasm Metastasis; Neoplasm Recurrence, Local
Keywords: Liver neoplasms; Liver metastases; MCRC; Litx™; LS11; Colorectal cancer with recurrent liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Neoplasm Recurrence, Local; Liver Neoplasms | interventions — Talaporfin; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Litx + Chemotherapy (Experimental)
  Interventions: Drug: Talaporfin sodium; Procedure: Percutaneous placement of device in liver metastases; Device: Interstitial light emitting diodes; Drug: FOLFOX4 regimen; Drug: FOLFIRI regimen
- Chemotherapy alone (Active Comparator)
  Interventions: Drug: FOLFOX4 regimen; Drug: FOLFIRI regimen

INTERVENTIONS:
Drug: Talaporfin sodium — LS11 (Talaporfin Sodium) dose is 1mg/kg administered intravenously slow push (3-5 minutes).
  Arms: Litx + Chemotherapy
Procedure: Percutaneous placement of device in liver metastases — Light Source placement will be conducted under placement imaging using ultrasound or CT guidance. No more than four Light Sources will be used at a single treatment session. The Light Sources may be used in a single lesion or in multiple lesions.
  Arms: Litx + Chemotherapy
Device: Interstitial light emitting diodes — 200 J/cm per Light Source at 20 mW/cm light energy
  Arms: Litx + Chemotherapy
Drug: FOLFOX4 regimen — Standard care chemotherapy regimen consisting of leucovorin, 5-FU and oxaliplatin
Drug: FOLFIRI regimen — Standard care chemotherapy regimen consisting of leucovorin, 5-FU and irinotecan

SUMMARY:
The purpose of the study is to assess the overall survival and progression free survival of patients treated with Litx™ + chemotherapy versus chemotherapy alone in the treatment of Colorectal Cancer with recurrent liver metastases, and to demonstrate the safety of Litx™ therapy.

Litx™ consists of a light-activated drug, talaporfin sodium (LS11, Light Sciences Oncology, Bellevue, Washington), and a light generating device, composed of light-emitting diodes (LEDs), that is energized by a power controller and percutaneously placed in the target tumor tissue inside the body.

DETAILED DESCRIPTION:
Randomized, stratified, two arm study:

* Litx™ and chemotherapy arm (FOLFOX4 or FOLFIRI)
* Chemotherapy only arm (FOLFOX4 or FOLFIRI)

For patients who have progressed on FOLFIRI, they will be treated with Litx™ plus FOLFOX4 versus FOLFOX4 alone; and for patients who have progressed on FOLFOX, they will be treated with Litx™ plus FOLFIRI versus FOLFIRI alone.

Stratification upon enrollment by chemotherapy and tumor sum of the longest diameter (SLD) (SLD < 4 cm or SLD ≥4 cm but ≤7.5 cm).

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent metastatic liver lesions from colorectal cancer who progressed on either FOLFOX or FOLFIRI
* Biopsy proven evidence of colorectal cancer
* At least one liver lesion that can be measured in one dimension at >10 mm with spiral CT scan (CT preferred but MRI allowed)
* ECOG Performance Status 0-2
* Life expectancy of at least 16 weeks
* At least 30 days must have elapsed since the completion of any prior antineoplastic therapy and the patient must have recovered from acute side effects before day 0
* Understanding and ability to sign written informed consent
* 18 years of age or more
* Adequate hematologic, liver and renal functions as evidenced by the following: WBC > 2.5 × 10^9/L ; Platelet Count > 100 × 10^9/L ; Hemoglobin > 90 g/L ; Neutrophils >1.5 × 10^9/L ; PT and PTT < 1.5 Control ; SGOT, SGPT < 5 × ULN ; GGT < 5 × ULN ; Alkaline phosphatase < 5 × ULN ; Bilirubin < 3 × ULN ; Creatinine < 1.5 × ULN

Exclusion Criteria:

* Patients who are candidates for complete surgical resection
* Patients who received bevacizumab (Avastin®) or cetuximab (Erbitux®) within 30 days of randomization. Use of bevacizumab or cetuximab is prohibited while participating in this study
* Patients who would require more than a total number of 12 light source applications over three Litx™ experimental treatments (no more than 4 light sources per treatment).
* Patients who have a single measurable tumor greater than 7.5 cm in any organ
* Target lesions irradiated within 3 months of randomization
* Patients with tumor involvement in greater than 50% of parenchyma of the liver
* Evidence of major vessel invasion of any organ
* Patients with any non-colorectal cancers except for adequately treated basal or squamous cell skin cancer, or adequately treated stage I or II cancer from which the patient has been disease-free for ≥ 3 years, or other cancer from which the patient has been disease-free for ≥ 5 years
* Known sensitivity to porphyrin-type drugs or known history of porphyria
* Pregnancy or breast-feeding patients. A negative pregnancy test (urine or serum) from women of childbearing age is required prior to enrollment. A fertile patient must use effective contraception during participation in the study
* Concurrent participation in another clinical trial involving experimental treatment
* Any concurrent disease or condition that in the opinion of the investigator impairs the patient's ability to complete the trial such as psychological, familial, sociological, geographical or medical conditions which in the Principal Investigator's opinion could compromise compliance with the objectives and procedures of this protocol or obscure interpretation of the trial's data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 483 (Actual)
Dates: Start 2007-02; Primary Completion 2011-05 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sy-Shi Wang, PhD, Study Director — Light Sciences Oncology
Locations (57):
- Austria (2):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Krankenhaus Hietzing mit Neurologischen Zentrum Rosenhugel, Vienna
- Bosnia and Herzegovina (2):
  - Clinical Hospital Mostar, Internal Clinic, Department of Gastroenterology, Mostar
  - Clinical Centre of the University of Sarajevo, Institute of Oncology, Sarajevo
- Croatia (4):
  - General Hospital Karlovac, Karlovac
  - Clinical Centre Zagreb, Clinical Oncology, Zagreb
  - General Hospital "Sveti Duh", Zagreb
  - University Hospital Dubrava, Zagreb
- Germany (5):
  - Ostalb-Klinikum Aalen Darmzentrum Medizinische Klinik I, Aalen
  - Helios Kliniken - Innere Medizin und Kardiologie, Borna
  - Katholisches Krankenhaus St. Johann Nepomuk, Erfurt
  - Johann Wolfgang Goethe Universitat, Frankfurt
  - Kliniken Ludwigsburg Bietigheim, Ludwigsburg
- India (8):
  - Bangalore Institute of Oncology, Bangalore, Karnataka
  - Mahavir Cancer Sansthan, Phulwarisharif, Patna
  - CIIGMA Institute of Medical Sciences, Aurangabad
  - Jawaharlal Nehru Cancer Hospital and Research Centre, Bhopal
  - SEAROC Cancer Center, S. K. Soni hospital, Jaipur
  - Shatabdi Super Specialty Hospital, Mumbai
  - Cancer Clinic, Shreevardhan complex, Nagpur
  - Ruby Hall Clinic, Pune
- Italy (4):
  - Azienda Ospedaliero-Universitaria Riunti, Ancona
  - Azienda Ospedaliera Careggi U.O. Oncologia Medica, Florence
  - Azienda Ospedaliera Universitaria Padovana, Padua
  - Policlinico Tor Vergata - Oncologia Medica, Rome
- Riga Eastern Hospital, Latvian Oncology Center, Riga, Latvia
- Poland (7):
  - Centrum Onkologii - Instytut im. Marii Skłodowskiej -Curie Oddział w Krakowie, Krakow
  - Szpital Uniwersytecki CMUJ, Klinika Chirurgii Ogólnej i Gastroenterologicznej, Krakow
  - Szpital Wojewódzki im. M. Kopernika, Klinika Chemioterapii Onkologicznej, Lodz
  - Klinika Chirurgii Onkologicznej, Lublin
  - Zakład Opieki Zdrowotnej MSWiA z Warmińsko-Mazurskim Centrum Onkologii, Olsztyn
  - Klinika Chirurgii Ogólnej i Onkologicznej, Szczecin
  - Centrum Onkologii - Instytut im. Marii Skłodowskiej -Curie, Klinika Nowotworów Jelita Grubego, Warsaw
- Romania (3):
  - Fundeni Clinical Institute, Bucharest
  - Oncology Institute "Ion Chircuta", Cluj-Napoca
  - St. Spiridon University Emergency Hospital, Iași
- Russia (11):
  - State Institution "Altay" Territorial Oncological Dispensary, Barmaul
  - Main Military Clinical Hospital named after Burdenko attached to Ministry of Defense of Russian Federation, Moscow
  - Municipal Cliical Hospital # 33 named after Ostroumov, Moscow
  - Russian Oncological Scientific Center named after Blokhin, Moscow
  - Privolzhsky District Medical Center, Nizhny Novgorod
  - Central Research Institute of Roentgenology and Radiology, Saint Petersburg
  - Scientific Research Institution of Oncology, Saint Petersburg
  - State Educational Institution of High Professional Education "Military-Medical Academy named after S.M. Kirov attached to Ministry of Defense of Russia", Saint Petersburg
  - Tambov Regional Oncological Dispensary, Tambov
  - State Healthcare Institution of Yaroslavl region, "Regional clinical oncological hospital", Yaroslavl
  - State Healthcare Institution "Sverdlovsk' Regional Oncological Dispensary", Yekaterinburg
- Serbia (3):
  - Institute of Oncology and Radiology of Serbia, Belgrade
  - Military Medical Academy, Belgrade
  - Institute of Oncology, Kamenitz
- Karolinska University Hospital, Stockholm, Sweden
- Ukraine (6):
  - Municipal Institution "Cherkassy" Regional Oncological Dispensary of Cherkassy, Cherkassy
  - Municipal Multiple-Discipline Clinical Hospital #4, Dnipro
  - Donetsk Cancer Centre, Donetsk
  - Kharkov Regional Clinical Oncology Dispansery, Kharkiv
  - The Central Hospital of the Ministry of Defense, Kyiv
  - Zaporozhye Medical Academy for postgraduate education, Zaporizhzhya

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Litx + Chemotherapy | Chemotherapy Alone
Started | 244 | 239
Treated | 222 | 232
Completed | 216 | 209
Not Completed | 28 | 30
Not completed — Lost to Follow-up | 4 | 5
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 15 | 14
Not completed — No Reply at EOS | 7 | 7
Not completed — Other | 1 | 0
Not completed — Status Unknown | 1 | 3

BASELINE CHARACTERISTICS:
Population: All patients randomized/enrolled
Groups:
- Total: Total of all reporting groups
Arm/Group | Litx + Chemotherapy | Chemotherapy Alone | Total
Number analyzed (Participants) | 244 | 239 | 483
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (9.8) | 60.1 (10.2) | 59.7 (10.0)
Age, Customized [Median (Full Range); unit: years] | 60.0 [20 to 83] | 61.0 [31 to 81] | 60.0 [20 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 97 | 204
  Male | 137 | 142 | 279

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Time from randomization to death
Time Frame: Up to 184 weeks
Population: ITT (All patient randomized/enrolled)
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Litx + Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 244 | 239
Days | 390 [234 to 735] | 405 [244 to 655]

ADVERSE EVENTS:
Arm/Group | Litx + Chemotherapy | Chemotherapy Alone
Serious Adverse Events (participants affected / at risk) | 66/222 | 52/232
Other Adverse Events (participants affected / at risk) | 201/222 | 207/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Litx + Chemotherapy (N=222) | Chemotherapy Alone (N=232)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 5 | 4
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 3 | 1
Bile duct obstruction (Hepatobiliary disorders) | 3 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Haemobilia (Hepatobiliary disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Liver abscess (Infections and infestations) | 2 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Malaria (Infections and infestations) | 1 | 0
Malignant tumour excision (Surgical and medical procedures) | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to perineum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 12
Neutropenia (Blood and lymphatic system disorders) | 6 | 6
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Perirectal abscess (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 8 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pyrexia (General disorders) | 4 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Renal failure acute (Renal and urinary disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Status epilepticus (Nervous system disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 1
Sudden death (General disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Litx + Chemotherapy (N=222) | Chemotherapy Alone (N=232)
Abdominal pain (Gastrointestinal disorders) | 39 | 37
Abdominal pain upper (Gastrointestinal disorders) | 8 | 5
Alanine aminotransferase increased (Investigations) | 3 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 11
Anaemia (Blood and lymphatic system disorders) | 34 | 35
Anxiety (Psychiatric disorders) | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 7
Asthenia (General disorders) | 33 | 44
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 9
Blood albumin decreased (Investigations) | 7 | 4
Blood alkaline phosphatase increased (Investigations) | 7 | 3
Blood pressure increased (Investigations) | 7 | 2
Catheterisation venous (Surgical and medical procedures) | 13 | 12
Chest pain (General disorders) | 3 | 5
Chills (General disorders) | 3 | 5
Constipation (Gastrointestinal disorders) | 15 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 10
Decreased appetite (Metabolism and nutrition disorders) | 24 | 20
Diarrhoea (Gastrointestinal disorders) | 40 | 46
Dizziness (Nervous system disorders) | 3 | 7
Dyspepsia (Gastrointestinal disorders) | 4 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Eastern cooperative oncology group performance status worsened (Investigations) | 10 | 7
Fatigue (General disorders) | 47 | 45
Gamma-glutamyltransferase increased (Investigations) | 7 | 5
Headache (Nervous system disorders) | 7 | 6
Hyperbilirubinaemia (Hepatobiliary disorders) | 6 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 5
Hypertension (Vascular disorders) | 14 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 6
Hypotension (Vascular disorders) | 0 | 8
Insomnia (Psychiatric disorders) | 8 | 11
Leukopenia (Blood and lymphatic system disorders) | 23 | 21
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Nausea (Gastrointestinal disorders) | 69 | 67
Neuropathy peripheral (Nervous system disorders) | 10 | 6
Neutropenia (Blood and lymphatic system disorders) | 48 | 43
Oedema peripheral (General disorders) | 12 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 6
Paraesthesia (Nervous system disorders) | 11 | 12
Peripheral sensory neuropathy (Nervous system disorders) | 10 | 19
Phlebitis (Vascular disorders) | 5 | 6
Procedural pain (Injury, poisoning and procedural complications) | 112 | 0
Pyrexia (General disorders) | 48 | 34
Red blood cell sedimentation rate increased (Investigations) | 1 | 5
Stomatitis (Gastrointestinal disorders) | 11 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 13
Urinary tract infection (Infections and infestations) | 8 | 8
Vomiting (Gastrointestinal disorders) | 37 | 40
Weight decreased (Investigations) | 13 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days